CLINICAL TRIAL: NCT01226758
Title: A Randomised Double-blind, Placebo-controlled, Phase 1b Trial to Evaluate the Safety, Tolerability and Protective Efficacy of the Influenza Vaccine Candidate, FLU-v, in an Influenza Challenge Model
Brief Title: Influenza Vaccine Challenge Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PepTcell Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLU-v-002
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Influenza
Keywords: Safety; Tolerability; Efficacy; Influenza; Flu; Virus; Vaccine
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FLU-v with adjuvant (Experimental)
  Interventions: Biological: Influenza vaccine (FLU-v)
- Placebo (Placebo Comparator): Adjuvant only placebo
  Interventions: Biological: Placebo (adjuvant only)

INTERVENTIONS:
Biological: Influenza vaccine (FLU-v) — FLU-v (sterile lyophilised mixture of polypeptide T-cell epitope sequences) and adjuvant. Administered by single subcutaneous injection.
  Arms: FLU-v with adjuvant
Biological: Placebo (adjuvant only) — Single subcutaneous injection of adjuvant
  Arms: Placebo

SUMMARY:
The purpose of this research is to study the safety, tolerability and effectiveness of the investigational influenza vaccine in healthy volunteers infected with an attenuated influenza A virus.

DETAILED DESCRIPTION:
The investigational influenza vaccine (FLU-v) contains multiple highly conserved T cell epitopes that are present on most influenza viruses, which have been identified as reactive in different human leukocyte antigen (HLA) populations; thus making it unlikely that anybody in the vaccinated population would be unable to mount an immune response to at least one of the epitopes contained in the vaccine.

In this study up to 44 will be vaccinated with the FLU-v experimental vaccine or a placebo in a 1:1 ratio. Volunteers will attend a screening visit, a vaccination visit, a 10-11 day overnight stay in a quarantine facility, and a follow-up visit to the P1 clinic.

Three weeks after being vaccinated with FLU-v or placebo, 30 volunteers will be taken to a Quarantine Unit to be exposed to the attenuated H3N2 study virus and then monitored by study physicians and nurses for a 10-11 day period. The other 14 volunteers will be held in reserve as back-ups. If fewer than 30 of the volunteers who travel to the Quarantine Unit are eligible to be exposed to the study virus, then volunteers who have been kept in reserve will be used.

Following discharge from the Quarantine Unit, volunteers will attend one study follow-up visit, 28 days after exposure to the study virus. Assessments will take place and samples will be taken from volunteers.

ELIGIBILITY:
Inclusion Criteria:

* General good health determined by a screening evaluation ≤120 days prior to IMP administration and on the day of admittance to quarantine
* Using methods of contraception, (e.g. spermicidal gel plus condom) for the entire duration of the study, up to the Study Completion visit, and refrain from fathering a child in the three months following study drug administration.
* Negative HIV, hepatitis B and C antibody screens
* Negative class A drugs, alcohol and nicotine screen
* Seronegative (≤10 HAI) for challenge virus
* Have not been vaccinated for influenza virus since 2006 (as determined in the medical history) or had a known influenza-like illness in the current season, defined as in the last 12 months

Exclusion Criteria:

* Presence of any significant acute or chronic, uncontrolled medical or psychiatric illness, including but not exclusive to the conditions listed in Appendix 2, that in the view of the Investigator is associated with increased risk of complications of respiratory viral illness
* Abnormal pulmonary function as evidenced by clinically significant abnormalities in spirometry
* Presence of household member or close contact who is: less than 3 years of age; known immunodeficient; receiving immunosuppressants; undergoing/soon to undergo chemotherapy; diagnosed with emphysema or COPD; is elderly residing in a nursing home; severe lung disease or medical condition; received a transplant (bone marrow or solid organ)
* History of asthma, COPD, pulmonary hypertension, reactive airway disease, or any chronic lung condition of any aetiology
* Any laboratory test or ECG which is abnormal and deemed by the investigator to be clinically significant
* Venous access inadequate for phlebotomy demands
* Regular daily smokers during the 6 months prior to study entry or those who have a significant history of any tobacco use at any time
* Subject is diabetic
* History or evidence of autoimmune disease or known impaired immune responsiveness
* Recent and/or recurrent history of autonomic dysfunction
* Receipt of systemic glucocorticoids, antiviral drugs, immunoglobulins or blood transfusions within 1 month, or any other cytotoxic or immunosuppressive drug within 6 months prior to vaccination. Receipt of any systemic chemotherapy agent at any time
* Presence of any febrile illness or symptoms of upper or lower tract respiratory infection in the 28 days prior to viral inoculation
* Any anatomic or neurological abnormality impairing the gag reflex or associated with an increased risk of aspiration, or history suggestive of such a problem or any abnormality significantly altering the anatomy of the nose or nasopharynx
* Known IgA deficiency, immotile cilia syndrome, or Kartagener's syndrome
* Nasal or sinus surgery within 30 days prior to vaccination
* Significant history of seasonal hay fever or a seasonal allergic rhinitis (SAR), or perennial allergic rhinitis (PAR), or chronic nasal or sinus condition
* Acute and/or chronic use of any medication or other product for symptoms of rhinitis or nasal congestion or for any chronic nasopharyngeal complaint, or chronic use of any intranasal medication for any indication
* Use of any prescription drugs, herbal supplements, within 4 weeks prior to vaccine administration
* Receipt of any investigational drug within 3 months, or prior participation in a clinical trial of any influenza vaccine, medication or experimental Influenza viral challenge delivered directly to the respiratory tract within 1 year
* Previous exposure to the IMP or similar substance
* History of multiple and recurring allergies and/or adverse reaction to any components of the IMP and challenge virus preparation
* History of allergy or intolerance to the following drugs: oseltamivir or zanamivir.
* Allergic to gentamicin

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Day -21 to Day 28
  The primary safety endpoint for the vaccination phase of the study is the evaluation of all AEs occurring up to Day 28 (final follow-up). AE details will be collected by subject questioning and review of a subject self-assessment diary card (completed for Days -21 to -14) at the clinic visit on Day -2

SECONDARY OUTCOMES:
Safety of FLU-v | Days -21 to 28
  The Safety of FLU-v will be assessed by recording:
  Area under the curve (AUC) of composite symptom score in the 6 days after inoculation (Days 0 to 5 inclusive; Physical examination; Clinical chemistry, haematology and urinalysis; Vital signs (blood pressure (BP), heart rate (HR) and respiration rate (RR)); Electrocardiogram; Oral temperature; and Concomitant medications.
Post-innoculation symptoms | Days 0 to 28
  Exploratory Endpoints - Symptoms measured by:
  Time to peak of composite symptom score, duration, and time to resolution of composite score from peak; Peak severity symptom composite score in the 6 days after inoculation; Duration of upper respiratory infection (URI) symptoms after influenza viral inoculation; Occurrence of URI symptoms 1) with and 2) without fever; and occurrence of any influenza-like illness with or without fever.
Post-innoculation virology | 6 days following inoculation
  Exploratory endpoint - Virology will be measured by recording an analysing:
  Area under the curve (AUC) of influenza viral shedding in the 6 days after inoculation; Time to peak of influenza viral shedding, duration, and time to resolution of influenza viral shedding from peak; Peak of influenza viral shedding in the 6 days after inoculation.
Post-innoculation fever | Days -21 to 28
  Exploratory endpoint - Post-innoculation fever will be assessed by:
  Area under the curve (AUC)and peak of fever; Duration of fever, time to peak fever, and time from peak to resolution of fever; Occurrence and duration of clinical illness with and without documented fever; Total tissue count and total mucus weight; Total number of individual tissues and total mucous weights; and humoral and cell-mediated immune responses to vaccine, pre-influenza challenge.
Protective Efficacy (PE) | Day 1 to 5 post-viral challenge
  Protective Efficacy measured by the proportion of cases prevented by the vaccine relative to placebo (the difference in attack rate for placebo vaccinated minus FLU-v vaccinated subjects divided by the placebo vaccinated group attack rate).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gilbert, MBBCh, MICR, Principal Investigator — Retroscreen Virology Limited
Locations (1):
- Retroscreen Virology Limited, London, United Kingdom

REFERENCES:
- [Derived] Pleguezuelos O, Robinson S, Fernandez A, Stoloff GA, Caparros-Wanderley W. Meta-Analysis and Potential Role of Preexisting Heterosubtypic Cellular Immunity Based on Variations in Disease Severity Outcomes for Influenza Live Viral Challenges in Humans. Clin Vaccine Immunol. 2015 Aug;22(8):949-56. doi: 10.1128/CVI.00101-15. Epub 2015 Jun 17. PMID 26084515
- [Derived] Pleguezuelos O, Robinson S, Fernandez A, Stoloff GA, Mann A, Gilbert A, Balaratnam G, Wilkinson T, Lambkin-Williams R, Oxford J, Caparros-Wanderley W. A Synthetic Influenza Virus Vaccine Induces a Cellular Immune Response That Correlates with Reduction in Symptomatology and Virus Shedding in a Randomized Phase Ib Live-Virus Challenge in Humans. Clin Vaccine Immunol. 2015 Jul;22(7):828-35. doi: 10.1128/CVI.00098-15. Epub 2015 May 20. PMID 25994549